CLINICAL TRIAL: NCT02412670
Title: A Prospective Phase II Trial of Neoadjuvant Systemic Chemotherapy Followed by Extirpative Surgery for Patients With High Grade Upper Tract Urothelial Carcinoma
Brief Title: Chemotherapy Before Surgery in Treating Patients With High Grade Upper Urinary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA8141; NCI-2014-02267 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA8141 (Other: ECOG-ACRIN Cancer Research Group); EA8141 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: High Grade Upper Tract Urothelial Carcinoma
Keywords: carcinoma; drug therapy; nephroureterectomy; urinary tract; urothelium
MeSH Terms: conditions — Carcinoma | interventions — Methotrexate; merphos; Vinblastine; Doxorubicin; Cisplatin; Platinum; Gemcitabine; Carboplatin; pegfilgrastim; Nephroureterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (methotrexate, vinblastine, doxorubicin, cisplatin) (Experimental): Patients receive methotrexate IV over 2-3 minutes, vinblastine IV, doxorubicin hydrochloride IV, and cisplatin IV over 4 hours on day 1. Pegfilgrastim at 6 mg is given once 24-48 hours after completion of chemotherapy. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without metastatic disease undergo nephroureterectomy and lymph node dissection 21-60 days after completion of chemotherapy.
  Interventions: Drug: Methotrexate; Drug: Vinblastine; Drug: Doxorubicin; Drug: Cisplatin; Drug: Pegfilgrastim; Procedure: Nephroureterectomy
- Arm B (gemcitabine, carboplatin) (Experimental): Patients receive gemcitabine hydrochloride IV over 30-60 minutes on days 1 and 8 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without metastatic disease undergo nephroureterectomy and lymph node dissection 21-60 days after completion of chemotherapy.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Procedure: Nephroureterectomy

INTERVENTIONS:
Drug: Methotrexate — Given IV
  Other Names: Folex; abitrexate; mexate
  Arms: Arm A (methotrexate, vinblastine, doxorubicin, cisplatin)
Drug: Vinblastine — Given IV
  Other Names: vinblastine sulfate
  Arms: Arm A (methotrexate, vinblastine, doxorubicin, cisplatin)
Drug: Doxorubicin — Given IV
  Other Names: Adriamycin R; Rubex R; Adriamycin RDF R; Adriamycin PFS R; hydroxydaunorubicin; hydroxydaunomycin; ADR
  Arms: Arm A (methotrexate, vinblastine, doxorubicin, cisplatin)
Drug: Cisplatin — Given IV
  Other Names: Cisdiaminedichloroplatinum; Cis-diaminedichloroplatinum (II); diaminedichloroplatinum; cis-platinum; platinum; Platinol; Platinol-AQ; DDP; CDDP; DACP; NSC 119875
  Arms: Arm A (methotrexate, vinblastine, doxorubicin, cisplatin)
Drug: Gemcitabine — Given IV
  Other Names: 2'-Deoxy-2'; 2'-difluorocytidine monohydrochloride; Gemzar
  Arms: Arm B (gemcitabine, carboplatin)
Drug: Carboplatin — Given IV
  Other Names: Paraplatin
  Arms: Arm B (gemcitabine, carboplatin)
Drug: Pegfilgrastim — Administered subcutaneously
  Other Names: Neulasta
  Arms: Arm A (methotrexate, vinblastine, doxorubicin, cisplatin)
Procedure: Nephroureterectomy — Undergo nephroureterectomy and lymph node dissection

SUMMARY:
This phase II trial studies how well giving chemotherapy before surgery works in treating patients with aggressive upper urinary tract cancer. Drugs used in chemotherapy, such as methotrexate, vinblastine, doxorubicin hydrochloride, cisplatin, gemcitabine hydrochloride, and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Removing the affected upper urinary tract by surgery is the recommended treatment for upper urinary tract cancer, but can cause loss of kidney function and prevent patients from being able to receive chemotherapy after surgery. Giving chemotherapy before surgery, when the kidneys are working at their maximum, may allow less tissue to be removed during surgery and may be more effective in treating patients with high grade upper urinary tract cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the rate of complete pathologic response (pCR = pT0pN0) as assessed by standard pathologic review attained by neoadjuvant systemic chemotherapy and nephroureterectomy.

SECONDARY OBJECTIVES:

I. To evaluate the safety of neoadjuvant systemic chemotherapy in patients with upper tract urothelial carcinoma preceding nephroureterectomy.

II. To evaluate distant recurrence-free survival of patients treated with neoadjuvant systemic chemotherapy preceding nephroureterectomy.

III. To evaluate event-free survival of patients treated with neoadjuvant systemic chemotherapy preceding nephroureterectomy.

IV. To evaluate bladder cancer-free survival of patients treated with neoadjuvant systemic chemotherapy preceding nephroureterectomy.

V. To evaluate cancer specific survival of patients treated with neoadjuvant systemic chemotherapy preceding nephroureterectomy.

VI. To evaluate renal functional outcomes of patients treated with neoadjuvant systemic chemotherapy preceding nephroureterectomy.

TERTIARY OBJECTIVES:

I. To collect pre-treatment and post-treatment tumor tissue, peripheral blood mononuclear cell (PBMC), peripheral blood plasma, and urine specimens for potential evaluations of markers of chemotherapy response/resistance.

OUTLINE: Patients are assigned to 1 of 2 treatment arms based on baseline renal function.

ARM A (CREATININE CLEARANCE [CRCL] > 50): Patients receive methotrexate intravenously (IV) over 2-3 minutes, vinblastine IV, doxorubicin hydrochloride IV, and cisplatin IV over 4 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without metastatic disease undergo nephroureterectomy and lymph node dissection 21-60 days after completion of chemotherapy.

ARM B (30 =< CRCL <= 50): Patients receive gemcitabine hydrochloride IV over 30-60 minutes on days 1 and 8 and carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients without metastatic disease undergo nephroureterectomy and lymph node dissection 21-60 days after completion of chemotherapy.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have high grade upper tract urothelial carcinoma proven by one of the following:

  * Biopsy;
  * Urinary cytology with a 3-dimensional upper urinary tract mass on cross-sectional imaging; or
  * Urinary cytology and a mass visualized during upper urinary tract endoscopy
* Patients must have a creatinine clearance >= 30 ml/min as determined by Cockcroft-Gault calculation or 24-hour urine creatinine clearance measurement within 28 days of registration to be eligible for the study
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Patients must have a left ventricular ejection fraction (LVEF) >= 50% by (either multigated acquisition [MUGA] or 2-dimensional [2-D] echocardiogram) within 28 days of registration
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin (HgB) >= 9
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2 X institutional upper limit of normal (ULN)
* Bilirubin within institutional normal limits (or < 2.5 X the ULN for patients with Gilbert's disease)
* Patients with concomitant primaries of the bladder/urethra are allowed, as long as these sites are surgically resected and non-invasive cancers (< cT1N0)
* Patients may have a history of resectable urothelial cancer (including neoadjuvant chemotherapy) as long as patients meet one of the following:

  * pT0, Tis, or T1N0 and have no evidence of disease (NED) for more than 2 years from surgery or chemotherapy;
  * pT2-3aN0 and NED for more than 3 years from surgery or chemotherapy; or
  * > pT3b, or N+ and NED for more than 5 years from surgery or chemotherapy
* Women of childbearing potential and sexually active males must use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study

Exclusion Criteria:

* Evidence of metastatic disease or clinically enlarged lymph nodes on computed tomography (CT) or magnetic resonance imaging (MRI) of the abdomen and pelvis and CT chest obtained within 28 days of registration (a negative biopsy is required for lymph nodes > 1 cm in size to confirm lack of involvement); patients with lymph nodes > 1 cm in whom a biopsy is deemed not feasible are not eligible; patients with elevated alkaline phosphatase or suspicious bone pain should also undergo baseline bone scans to evaluate for bone metastasis
* Any component of small cell carcinoma; other variant histologies are permitted provided the predominant (>= 50%) subtype is urothelial carcinoma
* Peripheral neuropathy > grade 2
* History of allergy or hypersensitivity to methotrexate, vinblastine, doxorubicin (doxorubicin hydrochloride), cisplatin, gemcitabine (gemcitabine hydrochloride), carboplatin or filgrastim or pegfilgrastim
* Another active second malignancy other than non-melanoma skin cancers and biochemical relapsed prostate cancer; patients that have completed all necessary therapy and are considered to be at less than 30% risk of relapse are not considered to have an active second malignancy and are eligible for enrollment
* Prior systemic doxorubicin for patients who have creatinine clearance that meets >= 50 ml/min
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction in last 3 months, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known to have human immunodeficiency virus (HIV) or are on combination antiretroviral therapy
* Prior radiation therapy to >= 25% of the bone marrow for other diseases or prior systemic anthracycline therapy; prior intravesical anthracycline therapy for non-muscle invasive urothelial carcinoma of the bladder is permitted
* Pregnant or breast-feeding; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2022-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Margulis, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (134):
- United States (134):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Tulsa Cancer Institute, Tulsa, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology at Evangelical Community Hospital, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Aurora Cancer Care-Burlington, Burlington, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Aurora Advanced Healthcare Inc-Menomonee Falls, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Result] Margulis V, Puligandla M, Trabulsi EJ, Plimack ER, Kessler ER, Matin SF, Godoy G, Alva A, Hahn NM, Carducci MA, Hoffman-Censits J; Collaborators. Phase II Trial of Neoadjuvant Systemic Chemotherapy Followed by Extirpative Surgery in Patients with High Grade Upper Tract Urothelial Carcinoma. J Urol. 2020 Apr;203(4):690-698. doi: 10.1097/JU.0000000000000644. Epub 2019 Nov 8. PMID 31702432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on April 1, 2015 and accrued its first patient on August 27, 2015. Arm A reached its accrual and was closed on May 31, 2017. Arm B was closed due to slow accrual on January 5, 2018.
Period: Overall Study
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Started | 30 | 6
Eligible and Treated | 29 | 6
Completed | 23 | 5
Not Completed | 7 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only eligible and treated patients are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin) | Total
Number analyzed (Participants) | 29 | 6 | 35
Age, Continuous [Median (Full Range); unit: years] | 65 [40 to 84] | 75 [53 to 78] | 66 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 23 | 4 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 27 | 4 | 31
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 26 | 4 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response Rate
Description: Complete pathologic response is defined as pT0pN0 (no evidence of disease) as assessed by pathologic evaluation of nephrectomy/ureterectomy and any identifiable regional lymph nodes.
Time Frame: Assessed at nephroureterectomy or regional lymph node dissection (21-60 days from completion of chemotherapy; chemotherapy was administered for a total of 4 cycles; cycle length is 14 days and 21 days for arms A and B, respectively)
Population: Eligible and treated patients
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 29 | 6
proportion of participants | 0.103 [0.039 to 0.216] | 0.167 [0.017 to 0.51]

2. Secondary Outcome: Recurrence-free Survival
Description: Recurrence-free survival is defined as the time from the date of surgery to disease recurrence or death from any cause. Patients alive without documented recurrence will be censored at the date of last disease assessment.
Time Frame: Assessed every 3 months for 2 years; and every 6 months for 3-5 years
Population: Eligible and treated patients who underwent radical nephro-ureterectomy and were rendered disease-free
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 28 | 5
months | NA [NA to NA] — Median was not reached. The upper and lower limits of the 90% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 8.5 [3.3 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

3. Secondary Outcome: Event-free Survival
Description: Event-free survival is defined as the time from registration to the earliest occurrence of recurrence of any type, disease progression, new invasive primary cancer, or death from any cause. Disease progression will be assessed using RECIST 1.1. Disease progression is defined as appearance of one or more new lesions, unequivocal progression of existing non-target lesions, or at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Assessed every 3 months for 2 years, and every 6 months for 3-5 years
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 29 | 6
months | NA [NA to NA] — Median was not reached. The upper and lower limits of the 90% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 10.2 [7.1 to NA] — The upper limit of the 90% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

4. Secondary Outcome: Bladder Cancer-free Survival
Description: Bladder cancer-free survival was defined as the time from the date of surgery to the earlier of a return of bladder cancer or death from any cause. Patients alive without documented bladder cancer were censored at the date of last disease assessment.
Time Frame: Assessed every 3 months for 2 years, and every 6 months for 3-5 years
Population: Eligible and treated patients who underwent radical nephro-ureterectomy and were rendered disease-free
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 28 | 5
months | NA [NA to NA] — Median was not reached. The upper and lower limits of the 90% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment. | NA [NA to NA] — Median was not reached. The upper and lower limits of the 90% confidence interval were not calculable because an insufficient number of participants reached the event at the final time point for assessment.

5. Secondary Outcome: Cumulative Incidence of Cancer-specific Death at 24 Months
Description: Cancer-specific survival was defined as the time from registration to death due to cancer; deaths due to other causes are counted as competing events. Cancer-specific survival was analyzed using Gray's method and cumulative incidence of cancer-specific death at 24 months is reported.
Time Frame: Assessed every 3 months for 2 years
Population: Eligible and treated patients
Measure: Number (90% Confidence Interval); unit: proportion of patients died of cancer
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 29 | 6
proportion of patients died of cancer | 0.09 [0.02 to 0.21] | 0.20 [0.01 to 0.56]

6. Secondary Outcome: Proportion of Patients With Renal Insufficiency at Completion of Chemotherapy
Description: Renal insufficiency is defined as CrCl < 60 ml/min.
Time Frame: Assessed at completion of chemotherapy; at 8 weeks for Arm A and 12 weeks for Arm B
Population: All patients with chemotherapy
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 30 | 6
proportion of participants | 0.2 [0.091 to 0.357] | 0.833 [0.418 to 0.991]

7. Secondary Outcome: Proportion of Patients With Renal Insufficiency at Completion of Surgery
Description: Renal insufficiency is defined as CrCl < 60 ml/min.
Time Frame: Assessed at completion of surgery (21-60 days from completion of chemotherapy; chemotherapy was administered for a total of 4 cycles; cycle length is 14 days and 21 days for arms A and B, respectively)
Population: All patients who underwent radical nephro-ureterectomy
Measure: Number (90% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
Number analyzed (Participants) | 29 | 6
proportion of participants | 0.69 [0.521 to 0.828] | 0.833 [0.418 to 0.991]

ADVERSE EVENTS:
Time Frame: Assessed every 2 weeks for arm A and every 3 weeks for arm B while on treatment and for 30 days after the end of treatment up to 5 years
Description: Serious adverse events are defined as treatment-related adverse events of grade 3 or higher. Other adverse events are treatment-related adverse events not included in the serious adverse events.
Arm/Group | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) | Arm B (Gemcitabine, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 2/30 | 1/6
Serious Adverse Events (participants affected / at risk) | 7/30 | 3/6
Other Adverse Events (participants affected / at risk) | 30/30 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) (N=30) | Arm B (Gemcitabine, Carboplatin) (N=6)
Anemia (Blood and lymphatic system disorders) | 2 | 2
Fatigue (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 2 | 2
Investigations - Other, specify (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Methotrexate, Vinblastine, Doxorubicin, Cisplatin) (N=30) | Arm B (Gemcitabine, Carboplatin) (N=6)
Anemia (Blood and lymphatic system disorders) | 20 | 5
Fatigue (General disorders) | 22 | 5
Nausea (Gastrointestinal disorders) | 23 | 4
Vomiting (Gastrointestinal disorders) | 6 | 2
Creatinine increased (Investigations) | 11 | 2
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 9 | 3
White blood cell decreased (Investigations) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT02412670/Prot_SAP_000.pdf